CLINICAL TRIAL: NCT00300651
Title: Phase 3 Randomized Controlled Trial of Cognitive Behavioural Therapy for Patients With Schizophrenia
Brief Title: Trial of Cognitive Behavioral Therapy for Schizophrenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philipps University Marburg (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PhilippsU
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Last update posted 2006-03-09 (Estimated); Status verified 2006-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Delusional Disorder
Keywords: Cognitive Behavioral Therapy; Schizophrenia; Cognitive Biases; Efficacy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy

SUMMARY:
The following study addresses the hypothesis that cognitive-behavioral interventions will be effective in reducing positive and negative symptoms of schizophrenia under the conditions of the German health care system. It is also hypothesized that interventions designed to reduce delusions will reduce cognitive biases and dysfunctional self-concepts.

DETAILED DESCRIPTION:
Background: In spite of the proven effectiveness in a series of randomized controlled studies, cognitive-behavioural interventions for the treatment of symptoms of schizophrenia have been not yet been evaluated under the conditions of the German health care system. Additionally, it remains unclear which processes are responsible for reducing positive symptoms using CBT-interventions.

Hypothesis: The following study addresses the hypothesis that CBT will be effective in reducing positive and negative symptoms of schizophrenia. It is also hypothesized that CBT will reduce cognitive biases and dysfunctional self-concepts.

Method: 70 patients with a primary diagnosis of schizophrenia will be randomized to a CBT-treatment- and a waiting-list-control-group. CBT involves a formulation-based treatment of approximately 25 sessions by trained and supervised therapists plus standard care (psychiatric medical treatment) in an outpatient setting. Participants will be referred from cooperating psychiatrists. Patients randomized to the waiting-list condition take part in the assessment phase, then receive standard care alone for 12 weeks and are then offered CBT. The primary outcome measure will be the Positive and Negative Syndrome Scale. Additionally, depression, dysfunctional self-concepts and cognitive biases will be assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* persons with a primary diagnosis of schizophrenia, schizoaffective disorder, delusional disorder acute or in incomplete remission a value of at least 3 on delusions, P1, P3 or G9 in Positive and Negative Syndrome Scale

fluent in German language

Exclusion Criteria:

* severe organic brain disease

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2006-03; Study Completion 2009-08

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS)before and after treatment and at 1-year-follow-up

SECONDARY OUTCOMES:
Depression before and after treatment and at 1-year-follow-up
Dysfunctional Attitudes before and after treatment and at 1-year-follow-up
Cognitive biases (jumping to conclusions, attribution, theory of mind) before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tania M Lincoln, PhD, Principal Investigator — Philipps-Universität Marburg, Faculty of Psychology, Section for Clinical Psychology and Psychotherapy; Tania M Lincoln, PhD, Study Director — Philipps-Universität Marburg, Faculty of Psychology, Section for Clinical Psychology and Psychotherapy
Locations (1):
- Philipps-Universität, Marburg, Germany

REFERENCES:
- See also: Related Info — http://www.psychotherapie-ambulanz-marburg.de/FrameSets/fsForschung.html